CLINICAL TRIAL: NCT01611857
Title: A Phase I/II Trial of the c-Met Inhibitor, Tivantinib, in Combination With FOLFOX for the Treatment of Patients With Advanced Solid Tumors (Phase I) and Previously Untreated Metastatic Adenocarcinoma of the Distal Esophagus, Gastroesophageal (GE) Junction, or Stomach (Phase II)
Brief Title: Phase I/II Trial of Tivantinib With FOLFOX for the Treatment of Advanced Solid Tumors and Previously Untreated Metastatic Adenocarcinoma of the Distal Esophagus, Gastroesophageal Junction or Stomach
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GI 157
Record Dates: First submitted 2012-06-01; First posted 2012-06-05 (Estimated); Results first posted 2016-11-23 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-10

CONDITIONS: Malignant Solid Tumour; Gastroesophageal Cancer
Keywords: Advanced solid tumors; First-Line Metastatic GE cancer; c-Met Inhibitor; Tivantinib; FOLFOX
MeSH Terms: interventions — ARQ 197; Folfox protocol; Fluorouracil; Leucovorin; Oxaliplatin; Levoleucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Maximum Tolerated Dose (Experimental): Phase I trial of Tivantinib plus FOLFOX for the treatment of patients with advanced solid tumors followed by a Phase II portion for patients with first-line metastatic GE cancer.
  Interventions: Drug: Tivantinib; Drug: FOLFOX

INTERVENTIONS:
Drug: Tivantinib — Patients with advanced solid tumors will be treated with oral Tivantinib (120, 240, or 360 mg BID) daily for 14 days in cycles of 14 days.
  Other Names: ARQ 197
Drug: FOLFOX — The FOLFOX treatment regimen is started on Day 1 of each cycle and consists of 5-Fluorouracil (5-FU) 400 mg/m^2, 5-FU continuous IV 2400 mg/m^2 over 46 hours, leucovorin 400 mg/m^2 IV, and oxaliplatin 85 mg/m^2.
  Other Names: 5-FU; Leucovorin; Oxaliplatin; Levoleucovorin; 5-Fluorouracil

SUMMARY:
This study is a Phase I/II trial of Tivantinib plus FOLFOX for the treatment of patients with advanced solid tumors. In Phase I the Maximum Tolerated Dose (MTD) will be determined; in Phase II patients with first-line metastatic GE cancer will be treated at the MTD. It is hypothesized that the response rate (RR) will be improved from 45% to at least 65% under this regimen.

DETAILED DESCRIPTION:
This is a Phase I, open-label, non-randomized, dose-escalation study with a Phase II portion planned upon reaching the Maximum Tolerated Dose or recommended Phase II dose (RP2D). Phase I: The first cycle of the Phase I portion of the trial will be considered the Dose Limiting Toxicity evaluation period. Patients with advanced solid tumors will be treated with Tivantinib on Days 1 to 14 and with FOLFOX on Day 1. Following evaluation of the Dose Limiting Toxicities, doses will be escalated/reduced according to the protocol with 3 to 6 patients treated per dose level until the Maximum Tolerated Dose is determined.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy ≥12 weeks.
* Karnofsky performance status ≥70%
* Patients must have measurable disease per RECIST Version 1.1.
* Adequate hematologic function defined as:
* Absolute neutrophil count (ANC) ≥1500/μL
* Hemoglobin (Hgb) ≥9 g/dL (5.6 mmol/L)
* Platelets ≥100,000/uL
* Adequate liver function defined as:
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST <2.5 x the institutional upper limit of normal (ULN) or ≤5.0 x the institutional ULN in patients with liver metastases.
* Total bilirubin within normal limits (WNL) (or ≤1.5 x the institutional ULN in patients with liver metastases; or total bilirubin ≤3.0 x ULN with direct bilirubin within normal limits in patients with well documented Gilbert Syndrome).
* Serum creatinine <1.5 X ULN or calculated 24-hour creatinine clearance >40 mL/min.
* Patients who are on coumadin should have an international normalized ratio (INR) value within the therapeutic range (i.e., 2 to 3 x ULN). Patients who are on stable, chronic doses of coumadin are eligible.

PHASE I ONLY

•Patients must have histologically confirmed solid tumor malignancy that is metastatic or unresectable and for which standard therapy would include FOLFOX or for which standard curative or palliative measures do not exist or are no longer effective.

PHASE II ONLY

* Histologic documentation of adenocarcinoma of the esophagus, GE junction, or stomach.
* Metastatic GE cancer as documented by radiologic study or surgical evidence of metastatic disease.
* No prior chemotherapy for metastatic disease. Previous combined modality therapy for locally advanced disease is allowed if completed ≥6 months prior to recurrence (acceptable chemotherapy drugs include 5-FU, capecitabine, cisplatin, carboplatin, paclitaxel, oxaliplatin, and docetaxel).
* Prior radiation therapy is allowed. At least 4 weeks must have elapsed from completion of the radiation therapy and all signs of toxicity must have resolved.
* Prior adjuvant chemotherapy is allowed if completed ≥6 months prior to the documentation of metastatic disease.

Exclusion Criteria:

* Patients with known central nervous system (CNS) metastases may be enrolled, provided the metastases have undergone treatment, the patient is asymptomatic, and the patient does not require antiepileptic drugs or steroids as treatment for the CNS metastases.
* Patients with poorly controlled or clinically significant atherosclerotic vascular disease including New York Heart Association Grade 3 or greater congestive heart failure; unstable angina ; myocardial infarction, cardiovascular accident, transient ischemic accidents, angioplasty, cardiac or vascular stenting in the past 6 months; or ventricular arrhythmia requiring medication. Patients with previously diagnosed symptomatic bradycardia will be ineligible.
* Medical history of prolonged QT syndrome (>450 ms).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit safety or compliance with study requirements.
* History of hypersensitivity to active or inactive excipients of any component of treatment (5-FU, leucovorin, oxaliplatin, or Tivantinib), or known dipyrimidine dehydrogenase deficiency.
* Patients with evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation).
* Significant vascular disease (e.g., aortic aneurysm requiring surgical repair, or recent peripheral arterial thrombosis) ≤6 months prior to Day 1 of treatment.
* Any known positive test for human immunodeficiency virus, hepatitis C virus or acute or chronic hepatitis B infection.
* Mental condition that would prevent patient comprehension of the nature of, and risk associated with, the study.
* Use of any non-approved or investigational agent ≤28 days or 5 half-lives prior to administration of the first dose of study drug, whichever is shorter.
* Patients may not receive any other investigational or anti-cancer treatments while participating in this study.
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter drug absorption (e.g. active inflammatory bowel disease, uncontrolled nausea, vomiting, diarrhea, or malabsorption syndrome).
* Inability to swallow whole capsules.

PHASE I ONLY

•Patients who have had radiation therapy, hormonal therapy, biologic therapy, investigational agents, or chemotherapy for cancer within 28 days or 5 half-lives of the chemotherapy or biologic/targeted agents, whichever is shorter, prior to Day 1 of the study.

PHASE II ONLY

•Past or current history of neoplasm other than the entry diagnosis with the exception of treated non-melanoma skin cancer or carcinoma in situ of the cervix, or other cancers cured by local therapy alone and a disease free survival ≥5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-07; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johanna C Bendell, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (9):
- United States (9):
  - Yale University School of Medicine, New Haven, Connecticut
  - Florida Cancer Specialists-South, Fort Myers, Florida
  - Florida Cancer Specialists-Sarasota, Sarasota, Florida
  - Florida Cancer Specialists-North, St. Petersburg, Florida
  - Oklahoma University, Oklahoma City, Oklahoma
  - South Carolina Oncology Associates, Columbia, South Carolina
  - Tennessee Oncology - Chattanooga, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Center for Cancer and Blood Disorders, Fort Worth, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between January 2012 and March 2014, 49 patients were enrolled at multiple centers in the U.S. Fifteen patients with advanced solid tumors were enrolled in the dose escalation phase, and 34 patients with first-line metastatic cancer of the esophagus, gastroesophageal (GE) junction, or stomach in the expansion phase.
Pre-assignment Details: Forty-nine patients were enrolled; 47 were treated. Two participants withdrew prior to dosing. 15 participants were enrolled and treated in the dose escalation phase. 34 participants were enrolled in the dose expansion phase; however only 32 were treated. Patients continued treatment until disease progression or intolerable toxicity.
Groups:
- Tivantinib + FOLFOX Dose Escalation: Tivantinib: (120 mg; 240 mg; or 360 mg) orally, twice daily (PO BID) on Days 1-14 of each 2 week cycle;
  FOLFOX: [5-Fluorouracil (5-FU) 400 mg/m^2, 5-FU continuous IV 2400 mg/m^2 over 46 hours, leucovorin 400 mg/m^2 IV, and oxaliplatin 85 mg/m^2] on Day 1 each cycle.
- Tivantinib + FOLFOX Dose Expansion: Tivantinib: 360 mg PO BID on Days 1-14 of each 2-week cycle.
  FOLFOX: (5-FU 400 mg/m^2, 5-FU continuous IV 2400 mg/m^2 over 46 hours, leucovorin 400 mg/m^2 IV, and oxaliplatin 85 mg/m^2) on Day 1 of each 2-week cycle.
Period: Overall Study
Arm/Group | Tivantinib + FOLFOX Dose Escalation | Tivantinib + FOLFOX Dose Expansion
Started | 15 (Three dose levels of tivantinib (120 mg, 240 mg, and 360 mg) were evaluated to determine the MTD.) | 34
Tivantinib 120 mg | 5 | 0
Tivantinib 240 mg | 3 | 0
Tivantinib 360 mg | 7 | 32 (Two participants withdrew prior to receiving drug.)
Completed | 15 | 32
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: In the Tivantinib + FOLFOX Dose Expansion 34 patients were enrolled; only 32 were treated. Two dropped out prior to treatment. The Intent-to-Treat (ITT) population includes all 34 patients. Safety assessment was based on the population that received at least one dose of drug (N = 32); the efficacy assessments used the ITT population (N = 34).
Groups:
- Tivantinib+FOLFOX Dose Escalation: Tivantinib: (120 mg, 240 mg, or 360 mg) orally, twice daily on Days 1-14 of each 2 week cycle.
  FOLFOX: (5-FU 400 mg/m^2, 5-FU continuous IV 2400 mg/m^2 over 46 hours, leucovorin 400 mg/m^2 IV, and oxaliplatin 85 mg/m^2) on Day 1 each cycle.
- Tivantinib+FOLFOX Dose Expansion: Tivantinib: 360 mg PO BID on Days 1-14 of each 2-week cycle;
  FOLFOX: (5-FU 400 mg/m^2, 5-FU continuous IV 2400 mg/m^2 over 46 hours, leucovorin 400 mg/m^2 IV, and oxaliplatin 85 mg/m^2) on Day 1 of each 2-week cycle.
  Treatment continued until disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Tivantinib+FOLFOX Dose Escalation | Tivantinib+FOLFOX Dose Expansion | Total
Number analyzed (Participants) | 15 | 34 | 49
Age, Continuous [Median (Full Range); unit: years] | 62 [33 to 72] | 65 [34 to 88] | 63.5 [33 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 10 | 26 | 36
Region of Enrollment [Number; unit: participants]
  United States | 15 | 34 | 49
Tumor Type [Number; unit: participants] — Participants enrolled per tumor type.
  participants
    Colorectal | 7 | 0 | 7
    Esophageal | 4 | 14 | 18
    Pancreatic | 1 | 0 | 1
    GE Junction | 1 | 9 | 10
    Cholangiocarcinoma | 1 | 0 | 1
    Unknown primary | 1 | 0 | 1
    Gastric | 0 | 11 | 11
Karnofsky Performance Score [Number; unit: participants] — Karnofsky Score: 100 (no complaints), 90 (able to carry on normal activities, minor signs/symptoms of disease), 80 (normal activity with effort), 70 (care for self, unable to carry on normal activity or to do active work), 60 (requires occasional assistance, but able to care for most needs), 50 (requires considerable assistance and frequent medical care), 40 (disabled, requires special care and assistance), 30 (severely disabled, hospitalisation indicated though death not imminent), 20 (very sick, hospitalisation necessary, active supportive treatment necessary), 10 (moribund), 0 (dead).
  participants
    100 | 2 | 7 | 9
    90 | 3 | 18 | 21
    80 | 10 | 3 | 13
    70 | 0 | 5 | 5
    60 | 0 | 0 | 0
    50 | 0 | 0 | 0
    40 | 0 | 0 | 0
    30 | 0 | 0 | 0
    20 | 0 | 0 | 0
    10 | 0 | 0 | 0
    0 | 0 | 0 | 0
    Unknown | 0 | 1 | 1
Number of Participants with Prior Radiation Therapy [Number; unit: participants]
  Received Prior Radiation: Yes | 5 | 11 | 16
  Received Prior Radiation: No | 10 | 23 | 33

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Dose Limiting Toxicities (DLT) in Phase I Dose Escalation
Description: Using a standard 3+3 design participants were enrolled in dose-escalating cohorts to determine the maximum tolerated dose (MTD) of tivantinib when given with FOLFOX (5-FU 400 mg/m^2, continuous IV 5-FU 2400 mg/m^2 over 46 hours, leucovorin 400 mg/m^2 IV, and oxaliplatin 85 mg/m^2). MTD is defined as the highest dose level at which no more than 1 of 6 patients experiences a DLT, assessed by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.
Time Frame: 14 Days (1 cycle)
Population: Patients were assessed for DLT if they received at least 85% of the scheduled doses of study drugs in cycle 1. In the Tivantinib 120 mg cohort two participants were replaced due to missed drug. In the Tivantinib 360 mg cohort one patient was replaced due to an allergic reaction to oxaliplatin.
Measure: Number; unit: participants
Groups:
- Tivantinib 120 mg (PO BID) + FOLFOX: Tivantinib 120 mg given orally, twice daily (PO BID) on Days 1-14 of each 14-day cycle;
  FOLFOX: (5-FU 400 mg/m^2, 5-FU continuous IV 2400 mg/m^2 over 46 hours, leucovorin 400 mg/m^2 IV, and oxaliplatin 85 mg/m^2) on Day 1 each cycle.
- Tivantinib 240 mg (PO BID) + FOLFOX: Tivantinib 240 mg given orally, twice daily (PO BID) on Days 1-14 of each 14-day cycle;
  FOLFOX: (5-FU 400 mg/m^2, 5-FU continuous IV 2400 mg/m^2 over 46 hours, leucovorin 400 mg/m^2 IV, and oxaliplatin 85 mg/m^2) on Day 1 each cycle.
- Tivantinib 360 mg (PO BID) + FOLFOX: Tivantinib 360 mg given orally, twice daily (PO BID) on Days 1-14 of each 14-day cycle cycle;
  FOLFOX: (5-FU 400 mg/m^2, 5-FU continuous IV 2400 mg/m^2 over 46 hours, leucovorin 400 mg/m^2 IV, and oxaliplatin 85 mg/m^2) on Day 1 each cycle.
Arm/Group | Tivantinib 120 mg (PO BID) + FOLFOX | Tivantinib 240 mg (PO BID) + FOLFOX | Tivantinib 360 mg (PO BID) + FOLFOX
Number analyzed (Participants) | 3 | 3 | 6
participants | 0 | 0 | 1

2. Secondary Outcome: Progression Free Survival in Phase II Dose Expansion
Description: Defined as the time from first treatment until objective tumor progression or death from any cause. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: every 8 weeks until treatment discontinuation, projected 18 months and then every 3 months thereafter up to 5 years from start of treatment.
Population: The analysis was performed on an Intent-to-Treat basis (N = 34) for all participants in the Phase II portion of the study. Median follow-up was 15 months (3-21 months)
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Tivantinib + FOLFOX Dose Expansion: Tivantinib: 360 mg PO BID on Days 1-14 of each 14-day cycle. FOLFOX: (5-FU 400 mg/m^2, 5-FU continuous IV 2400 mg/m^2 over 46 hours, leucovorin 400 mg/m^2 IV, and oxaliplatin 85 mg/m^2) on Day 1 of each 14-day cycle.
  Treatment continued until disease progression or unacceptable toxicity.
Arm/Group | Tivantinib + FOLFOX Dose Expansion
Number analyzed (Participants) | 34
months | 6.1 [3.6 to 7.8]

3. Secondary Outcome: Overall Survival in Phase II Dose Expansion
Description: Defined as the time from first treatment until death from any cause.
Time Frame: every 8 weeks until treatment discontinuation, an expected average of 18 months, then every 12 weeks thereafter up to 5 years from start of treatment.
Population: The analysis was performed on an Intent-to-Treat basis (N=34) for all participants in the Phase II portion of the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tivantinib + FOLFOX Dose Expansion
Number analyzed (Participants) | 34
months | 9.6 [7.2 to NA] — The upper limit of the 95% Confidence Interval had not been reached at the time of analysis.

4. Secondary Outcome: Time to Progression in Phase II Dose Expansion
Description: Defined as the time from first treatment until objective tumor progression. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: every 8 weeks until progressive disease, expected 18 months.
Population: The analysis was performed on all participants (N = 34) in the Phase II portion of the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tivantinib + FOLFOX Dose Expansion
Number analyzed (Participants) | 34
months | 7.0 [5.7 to 11.5]

ADVERSE EVENTS:
Time Frame: Collected from day of first dose to 30 days after last dose of study medication up to 18 months.
Groups:
- Tivantinib+FOLFOX Dose Escalation: Tivantinib: orally, twice daily (PO BID) on Days 1-14 of each 2 week cycle; FOLFOX: (5-FU 400 mg/m^2, 5-FU continuous IV 2400 mg/m^2 over 46 hours, leucovorin 400 mg/m^2 IV, and oxaliplatin 85 mg/m^2) on Day 1 each cycle.
- Tivantinib+FOLFOX Dose Expansion: Tivantinib: 360 mg PO BID on Days 1-14 of each 2-week cycle. FOLFOX: (5-FU 400 mg/m^2, 5-FU continuous IV 2400 mg/m^2 over 46 hours, leucovorin 400 mg/m^2 IV, and oxaliplatin 85 mg/m^2) on Day 1 of each 2-week cycle.
  Treatment continued until disease progression or unacceptable toxicity.
Arm/Group | Tivantinib+FOLFOX Dose Escalation | Tivantinib+FOLFOX Dose Expansion
Serious Adverse Events (participants affected / at risk) | 6/15 | 17/32
Other Adverse Events (participants affected / at risk) | 14/15 | 31/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tivantinib+FOLFOX Dose Escalation (N=15) | Tivantinib+FOLFOX Dose Expansion (N=32)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Diarhhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Optic nerve disorder (Eye disorders) | 0 (0) | 1 (1)
Bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Ischemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tivantinib+FOLFOX Dose Escalation (N=15) | Tivantinib+FOLFOX Dose Expansion (N=32)
Neutropenia (Blood and lymphatic system disorders) | 4 (7) | 20 (20)
Fatigue (General disorders) | 8 (10) | 18 (18)
Nausea (Gastrointestinal disorders) | 7 (8) | 16 (16)
Diarrhea (Gastrointestinal disorders) | 5 (6) | 16 (16)
Peripheral neuropathy (Nervous system disorders) | 5 (10) | 14 (14)
Temperature intolerance (General disorders) | 1 (1) | 10 (10)
Mucositis (General disorders) | 0 (0) | 9 (9)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (14) | 9 (9)
Anemia (Blood and lymphatic system disorders) | 5 (14) | 8 (8)
Constipation (Gastrointestinal disorders) | 5 (5) | 8 (8)
Vomiting (Gastrointestinal disorders) | 3 (5) | 8 (8)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 6 (6)
Dizziness (Nervous system disorders) | 2 (2) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Asthenia (General disorders) | 0 (0) | 3 (3)
Bradycardia (Cardiac disorders) | 0 (0) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Weight decreased (Investigations) | 2 (2) | 3 (3)
Candida infection (Infections and infestations) | 0 (0) | 2 (2)
Chills (General disorders) | 2 (2) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 2 (2) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Edema (General disorders) | 1 (3) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Oral pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Paresthesia (Nervous system disorders) | 1 (2) | 2 (2)
Pyrexia (General disorders) | 2 (2) | 2 (2)
Visual impairment (Eye disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (2) | 1 (1)
Blood bilirubin increased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
QT prolongation (Investigations) | 3 (6) | 2 (5)
Proctolgia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (3)
Maculo-papular rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 1 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 3 (4)
Erythematous rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Muscosal inflammation (Gastrointestinal disorders) | 1 (1) | 6 (7)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral edema (General disorders) | 1 (1) | 0 (0)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.